CLINICAL TRIAL: NCT06073015
Title: Effect of Esketamine on Reducing Postoperative Anxiety and Depression in Adolescent Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: henanLYH
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Anxiety-depression
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Esketamine (0.25mg/kg)
  Interventions: Drug: Esketamine
- Control group (No Intervention): the same volume of normal saline

INTERVENTIONS:
Drug: Esketamine — Group S received a subanesthetic dose of esketamine 0.2mg/kg (2ml/50 mg) 5 minutes before the procedure began.
  Arms: Experimental group

SUMMARY:
This study intends to conduct a prospective, double-blind, randomized, controlled trial. Adolescents aged 8-17 years old are selected as subjects. Esketamine is used as intervention before surgery, vital signs data, serum IL-6, CRP and other inflammatory indicators are collected during surgery, and the incidence and degree of anxiety and depression are evaluated after surgery. To determine the effect of esketamine on reducing anxiety and depression in adolescents after surgery, and to provide an effective clinical basis for accelerating the rehabilitation of adolescents after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 8 years ≤ age ≤17 years;
2. Patients who plan to undergo elective surgery under general anesthesia, and the operation time is ≥2h;
3. ASA grade I-II

Exclusion Criteria:

1. Patients expected to be admitted to ICU after surgery;
2. Patients who need to return to the ward with tracheal intubation after surgery;
3. Allergic to the active ingredients or excipients of isketamine hydrochloride injection;
4. Patients with severe consciousness disorder or mental system disease (schizophrenia, mania, bipolar disorder, psychosis, etc.) or cognitive dysfunction;
5. Patients with congenital heart disease and severe developmental delay;
6. Patients with one of the following contraindications to esketamine :(a) patients at risk of a significant increase in blood pressure or intracranial pressure; (b) Patients with ocular hypertension (glaucoma) or penetrating ocular trauma; (c) Patients with poorly controlled or untreated hypertension (resting systolic blood pressure greater than 180 mmHg or resting diastolic blood pressure greater than 100 mmHg); (d) Untreated or undertreated hyperthyroidism;
7. Previous history of ketamine abuse or dependence, drug or alcohol dependence for more than 6 months, previous ketamine ineffective tests or adverse reactions.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depression scale scores 1 month after surgery | 1 month
  Anxiety and depression scale scores 1 month after surgery